CLINICAL TRIAL: NCT06714552
Title: Effect of the Replacement of Glycaemic Carbohydrates With Galacto-Oligosaccharide (GOS) Supplementation on Postprandial Glycaemic Response in Healthy Adults
Brief Title: Effect of a Sugar Replacement on Blood Glucose Levels in Healthy Adults
Acronym: SURE-BloG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Collaborators: Yakult Honsha Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: SURE-BloG
Record Dates: First submitted 2024-11-21; First posted 2024-12-03 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Postprandial Hyperglycemia; Hyperinsulinemia
Keywords: galacto-oligosaccharides; postprandial glycaemia; GOS
MeSH Terms: conditions — Hyperglycemia; Hyperinsulinism | interventions — 4'-galactooligosaccharide; Glucose

STUDY DESIGN:
Who Masked: Participant
Masking Description: Statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beta-galacto-oligosaccharide (Experimental)
  Interventions: Dietary Supplement: Galacto-Oligosaccharide
- Glucose (Other): Control
  Interventions: Other: Glucose

INTERVENTIONS:
Dietary Supplement: Galacto-Oligosaccharide — 24.0 g Oligomate® in 100 mL water
  Arms: Beta-galacto-oligosaccharide
Other: Glucose — 17.8 g glucose in 100 mL water
  Arms: Glucose

SUMMARY:
Diabetes and cardiovascular disease account for millions of deaths per year. One of the risk factors for both conditions is high blood sugar, particularly after eating (postprandial hyperglycaemia). Lowering blood sugar levels after a meal is expected to have a positive effect on preventing metabolic and cardiovascular diseases and improving the metabolic control of those who already suffer from these conditions.

The aim of this study is to investigate the effect of Oligomate® (beta-galacto-oligosaccharide) on postprandial glycaemia when used as a partial replacement of glycaemic carbohydrates in a beverage in otherwise healthy volunteers. Volunteers will be given water with either Oligomate® or glucose (control) added. Blood samples will be collected at eight time points (two before drinking the beverage and six after) to measure glucose and insulin levels.

DETAILED DESCRIPTION:
A single-centre, single-blind, randomised, controlled, cross-over, acute feeding trial will be conducted. The recruitment and study visits will be carried out at the Human Intervention Studies Unit (HISU) of the Rowett Institute.

A recruitment visit will be scheduled to screen for eligibility. During the visit, informed consent will be obtained before volunteers complete a health questionnaire, have their height and weight measured, and their veins checked to assess suitability for blood sample collection. A finger prick blood sample will then be taken to measure HbA1c levels. If a volunteer is eligible, the first study visit will be scheduled and they will be asked to fast for 12 hours the night before. A frozen high carbohydrate vegetarian ready-meal will be provided, which they will consume at home the evening before the study visit and before the fasting period.

During the study visits, the postprandial glycaemic response will be measured immediately after consumption of the supplement or control on two occasions separated by a wash-out period of 7-14 days. Briefly, subjects will arrive in the morning after having consumed the high carbohydrate meal the night before, followed by a 12 hr overnight fast. After recording body weight, a cannula will be inserted into an antecubital vein of one arm by a trained cannulist to allow repeated blood sampling during the assessment (approx. 6 ml collected per sample time to a total of 48 ml per visit). After obtaining two initial fasting blood samples (at -10min and -5min), subjects will consume the test beverage within 5 min. Further blood samples will be obtained at 15, 30, 45, 60, 90 and 120 min after ingestion to complete the postprandial glycaemic response assessment.

At the end of the first visit volunteers will receive the second ready-meal, identical to the first, which they will be asked to consume the evening before the second study visit, before the fasting period commences. During the second study visit, participants will consume the same beverage with the alternate supplement and complete the opposite arm of the postprandial glycaemic response assessment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Men or Women
* Body Mass Index (BMI) 18.5-29.9 kg/m^2
* Between 18 and 65 years of age
* Compliant (i.e., understands and is willing, able, and likely to comply with the experimental procedure and safety guidelines)
* Able to provide informed consent
* Premenopausal women must have a regular cycle or be on hormonal contraception.

Exclusion Criteria:

* Diabetes mellitus (all types including gestational diabetes)
* HbA1c result over the study limit [healthy range of between 4% and 5.9%]
* Endocrine disease (e.g., Cushing's syndrome)
* Any food allergy or intolerance, or following Vegan diet
* Medications that increase blood glucose (e.g., steroids, protease inhibitors, antipsychotics, antihypertensives, statins, diuretics, nicotinic acid, etc.)
* Medications that lower glycemia (e.g., anti-hyperglycaemics, insulin, beta- blockers, etc.)
* Medication affecting glucose regulation, appetite, and/or digestion/absorption of nutrients, antibiotics
* Major medical or surgical event requiring hospitalization in the previous 3 months
* Pregnant or lactating
* Participation in another clinical/supplementation trial or actively trying to reduce body weight
* Unable to comply with experimental procedures and safety guidelines
* Unable to give consent
* Smokers
* Travel during the study period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Difference in plasma glucose incremental area under the curve (iAUC) between study arms | 10 and 5 min before beverage consumption, 15, 30, 45, 60, 90, 120 min after beverage consumption
  Plasma glucose levels obtained from blood samples collected before and after beverage consumption will be determined using an automated clinical analyser. iAUC will be calculated using the trapezoidal rule with the baseline value of fasting plasma glucose subtracted.

SECONDARY OUTCOMES:
Difference in plasma glucose total area under the curve (tAUC) between study arms | 10 and 5 min before beverage consumption, 15, 30, 45, 60, 90, 120 min after beverage consumption
  Plasma glucose levels obtained from blood samples collected before and after beverage consumption will be determined using an automated clinical analyser. tAUC will be calculated using the trapezoidal rule with zero as the baseline.
Difference in peak plasma glucose concentration between study arms | 10 and 5 min before beverage consumption, 15, 30, 45, 60, 90, 120 min after beverage consumption
  Plasma glucose levels obtained from blood samples collected before and after beverage consumption will be determined using an automated clinical analyser. The peak plasma glucose concentrations for each arm will be compared.
Measured maximal incremental glucose value (iCMax) between study arms | 10 and 5 min before beverage consumption, 15, 30, 45, 60, 90, 120 min after beverage consumption
  Plasma glucose levels obtained from blood samples collected before and after beverage consumption will be determined using an automated clinical analyser. iCMax will be calculated using fasting plasma glucose levels as baseline.
Difference in plasma insulin iAUC between study arms | baseline, 30, 60, 120 min after beverage consumption
  Plasma insulin levels will be determined using ELISA from blood samples obtained, at several time points.
  iAUC will be calculated using the trapezoidal rule with baseline value of fasting plasma insulin subtracted.
Difference in plasma insulin tAUC between study arms | baseline, 30, 60, 120 min after beverage consumption
  Plasma insulin levels will be determined using ELISA from blood samples obtained at several time points. tAUC will be calculated using the trapezoidal rule with zero as the baseline.
Difference in peak plasma insulin concentration between study arms | baseline, 30, 60, 120 min after beverage consumption
  Plasma insulin will be determined using ELISA from blood samples obtained at several time points. Peak plasma insulin levels for each arm will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Scott, PhD, Principal Investigator — University of Aberdeen
Locations (1):
- University of Aberdeen, Rowett Institute, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The study is designed to look at average responses to the supplement. There is no need to share individual participant data.

REFERENCES:
- [Background] Venn BJ, Green TJ. Glycemic index and glycemic load: measurement issues and their effect on diet-disease relationships. Eur J Clin Nutr. 2007 Dec;61 Suppl 1:S122-31. doi: 10.1038/sj.ejcn.1602942. PMID 17992183
- [Background] Wright E Jr, Scism-Bacon JL, Glass LC. Oxidative stress in type 2 diabetes: the role of fasting and postprandial glycaemia. Int J Clin Pract. 2006 Mar;60(3):308-14. doi: 10.1111/j.1368-5031.2006.00825.x. PMID 16494646
- [Background] Blaak EE, Antoine JM, Benton D, Bjorck I, Bozzetto L, Brouns F, Diamant M, Dye L, Hulshof T, Holst JJ, Lamport DJ, Laville M, Lawton CL, Meheust A, Nilson A, Normand S, Rivellese AA, Theis S, Torekov SS, Vinoy S. Impact of postprandial glycaemia on health and prevention of disease. Obes Rev. 2012 Oct;13(10):923-84. doi: 10.1111/j.1467-789X.2012.01011.x. Epub 2012 Jul 11. PMID 22780564
- [Background] Neri S, Calvagno S, Mauceri B, Misseri M, Tsami A, Vecchio C, Mastrosimone G, Di Pino A, Maiorca D, Judica A, Romano G, Rizzotto A, Signorelli SS. Effects of antioxidants on postprandial oxidative stress and endothelial dysfunction in subjects with impaired glucose tolerance and type 2 diabetes. Eur J Nutr. 2010 Oct;49(7):409-16. doi: 10.1007/s00394-010-0099-6. Epub 2010 Mar 7. PMID 20213326
- [Background] Bonora E. Postprandial peaks as a risk factor for cardiovascular disease: epidemiological perspectives. Int J Clin Pract Suppl. 2002 Jul;(129):5-11. PMID 12166607
- [Background] Levitan EB, Song Y, Ford ES, Liu S. Is nondiabetic hyperglycemia a risk factor for cardiovascular disease? A meta-analysis of prospective studies. Arch Intern Med. 2004 Oct 25;164(19):2147-55. doi: 10.1001/archinte.164.19.2147. PMID 15505129
- [Background] Lin PJ, Borer KT. Third Exposure to a Reduced Carbohydrate Meal Lowers Evening Postprandial Insulin and GIP Responses and HOMA-IR Estimate of Insulin Resistance. PLoS One. 2016 Oct 31;11(10):e0165378. doi: 10.1371/journal.pone.0165378. eCollection 2016. PMID 27798656
- [Background] Hinnen DA. Therapeutic Options for the Management of Postprandial Glucose in Patients With Type 2 Diabetes on Basal Insulin. Clin Diabetes. 2015 Oct;33(4):175-80. doi: 10.2337/diaclin.33.4.175. PMID 26487791
- [Background] Kamruzzaman M, Horowitz M, Jones KL, Marathe CS. Gut-Based Strategies to Reduce Postprandial Glycaemia in Type 2 Diabetes. Front Endocrinol (Lausanne). 2021 Apr 9;12:661877. doi: 10.3389/fendo.2021.661877. eCollection 2021. PMID 33897622
- [Background] Gill SK, Rossi M, Bajka B, Whelan K. Dietary fibre in gastrointestinal health and disease. Nat Rev Gastroenterol Hepatol. 2021 Feb;18(2):101-116. doi: 10.1038/s41575-020-00375-4. Epub 2020 Nov 18. PMID 33208922
- [Background] Jenkins DJ, Goff DV, Leeds AR, Alberti KG, Wolever TM, Gassull MA, Hockaday TD. Unabsorbable carbohydrates and diabetes: Decreased post-prandial hyperglycaemia. Lancet. 1976 Jul 24;2(7978):172-4. doi: 10.1016/s0140-6736(76)92346-1. PMID 73796
- [Background] Bonsu NKA, Johnson S. Effects of inulin fibre supplementation on serum glucose and lipid concentration in patients with type 2 diabetes. International Journal of Diabetes and Metabolism. 2012 12;20(3):80-6. doi: 10.1159/000497730.
- [Background] Dehghan P, Pourghassem Gargari B, Asgharijafarabadi M. Effects of high performance inulin supplementation on glycemic status and lipid profile in women with type 2 diabetes: a randomized, placebo-controlled clinical trial. Health Promot Perspect. 2013 Jun 30;3(1):55-63. doi: 10.5681/hpp.2013.007. eCollection 2013. PMID 24688953
- [Background] Luo J, Van Yperselle M, Rizkalla SW, Rossi F, Bornet FR, Slama G. Chronic consumption of short-chain fructooligosaccharides does not affect basal hepatic glucose production or insulin resistance in type 2 diabetics. J Nutr. 2000 Jun;130(6):1572-7. doi: 10.1093/jn/130.6.1572. PMID 10827212
- [Background] Gargari BP, Namazi N, Khalili M, Sarmadi B, Jafarabadi MA, Dehghan P. Is there any place for resistant starch, as alimentary prebiotic, for patients with type 2 diabetes? Complement Ther Med. 2015 Dec;23(6):810-5. doi: 10.1016/j.ctim.2015.09.005. Epub 2015 Sep 16. PMID 26645521
- [Background] Liu F, Li P, Chen M, Luo Y, Prabhakar M, Zheng H, He Y, Qi Q, Long H, Zhang Y, Sheng H, Zhou H. Fructooligosaccharide (FOS) and Galactooligosaccharide (GOS) Increase Bifidobacterium but Reduce Butyrate Producing Bacteria with Adverse Glycemic Metabolism in healthy young population. Sci Rep. 2017 Sep 18;7(1):11789. doi: 10.1038/s41598-017-10722-2. PMID 28924143
- [Background] Muller M, Hermes GDA, Emanuel E C, Holst JJ, Zoetendal EG, Smidt H, Troost F, Schaap FG, Damink SO, Jocken JWE, Lenaerts K, Masclee AAM, Blaak EE. Effect of wheat bran derived prebiotic supplementation on gastrointestinal transit, gut microbiota, and metabolic health: a randomized controlled trial in healthy adults with a slow gut transit. Gut Microbes. 2020 Nov 9;12(1):1704141. doi: 10.1080/19490976.2019.1704141. Epub 2020 Jan 25. PMID 31983281
- [Background] Lightowler H, Thondre S, Holz A, Theis S. Replacement of glycaemic carbohydrates by inulin-type fructans from chicory (oligofructose, inulin) reduces the postprandial blood glucose and insulin response to foods: report of two double-blind, randomized, controlled trials. Eur J Nutr. 2018 Apr;57(3):1259-1268. doi: 10.1007/s00394-017-1409-z. Epub 2017 Mar 3. PMID 28255654
- See also: Indicator Metadata Registry List: Mean fasting blood glucose — https://www.who.int/data/gho/indicator-metadata-registry/imr-details/2380
- See also: Noncommunicable diseases — https://www.who.int/news-room/fact-sheets/detail/noncommunicable-diseases